CLINICAL TRIAL: NCT00694278
Title: Clinical Evaluation of the Effect of Duodenal-Jejunal Bypass on Type 2 Diabetes in Adults
Brief Title: Clinical Evaluation of the Effect of Duodenal-Jejunal Bypass on Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ferzli, George S., M.D. F.A.C.S. (Individual)
Responsible Party: Georger Ferzli M.D F.A.C.S., Lutheran Medical Center
Other Study IDs: LMC95
Record Dates: First submitted 2008-06-05; First posted 2008-06-10 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
The aim of this study and the primary outcome is to clinically evaluate effect of laparoscopic duodenal-jejunal bypass on non-obese type 2 diabetes. Secondary outcomes will evaluate CCK, FFA, Cholesterol Ghrelin, C-peptide, and HbA1c levels. Patients will be followed closely to ensure the desired results are sustained in long term

ELIGIBILITY:
Inclusion Criteria:

* Adults age 20-65 years
* Clinical diagnosis of type II diabetes buy on of the following three criteria (American Diabetes Association)

  1. A normal or high C-peptide level (to exclude type 1 diabetes) (>.9ng/ml)
  2. A random plasma glucose of 200mg/dl or more with typical symptom of diabetes
  3. A fasting plasma glucose of 126mg/dl or more on more than one occasion
* BMI 22-34 KG/m2
* Patients on oral hypoglycemic medications or insulin to control T2DM
* Inadequate control of diabetes as defined as HbA1c>7.5
* No contraindication for surgery or General Anesthesia as determined by multidisciplinary surgical team
* Ability to understand and describe the mechanism of action of ricks and benefits of the operation

Exclusion Criteria:

* Patients who meet any of the following exclusion criteria will be exclusion criteria will be excluded from enrollment into the study
* Enrolled in another clinical study which involves and investigational drug
* Diagnosis type 1 diabetes
* Pregnancy (all female patients will have beta HCG) or planned pregnancy within 2 years of entry into the study or unwilling to use reliable contraceptive method
* Previous gastric or esophageal surgery
* Immunosuppressive drugs including corticosteroids
* Coagulopathy (INR>1.5 or platelets<50,000/ul)
* Anemia (Hgb<10.0g/dl)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care office
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2008-06

CONTACTS AND LOCATIONS:
Overall Officials: George Ferzli, MD, Study Chair — Lutheran Medical Center
Locations (1):
- Lutheran Medical Center, Brooklyn, New York, United States